CLINICAL TRIAL: NCT03370874
Title: Phase 3 Clinical Study to Evaluate Efficacy and Safety of ALLO-ASC-DFU in Patients With Diabetic Foot Ulcers: A Randomized, Placebo-controlled, Double-blind, Parallel-group, Multi-center Study
Brief Title: Clinical Study to Evaluate Efficacy and Safety of ALLO-ASC-DFU in Patients With Diabetic Foot Ulcers.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALLO-ASC-DFU-301
Record Dates: First submitted 2017-11-28; First posted 2017-12-13 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALLO-ASC-DFU (Experimental): Hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells
  Interventions: Biological: ALLO-ASC-DFU
- Vehicle Sheet (Placebo Comparator): Hydrogel sheet without Allogenic mesenchymal stem cell
  Interventions: Procedure: Vehicle sheet

INTERVENTIONS:
Biological: ALLO-ASC-DFU — Application of ALLO-ASC-DFU sheet to diabetic foot ulcer
  Other Names: Hydrogel sheet containing allogenic mesenchymal stem cells
  Arms: ALLO-ASC-DFU
Procedure: Vehicle sheet — Application of Vehicle sheet to diabetic foot ulcer
  Other Names: Hydrogel sheet without Allogenic mesenchymal stem cell
  Arms: Vehicle Sheet

SUMMARY:
This is a phase III double-blind study to evaluate the efficacy and safety of ALLO-ASC-DFU in patients with Diabetic Foot Ulcer, compared to placebo therapy.

DETAILED DESCRIPTION:
Experimental: ALLO-ASC-DFU, Placebo Comparator: Vehicle Sheet, Study type: Interventional, Study design: Randomized, Placebo-controlled, Double-blind, Parallel-group, Multi-center Study

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18 and 75 years of age.
2. Subject is diagnosed with Type I or Type II diabetics and has diabetic foot ulcers for longer than 4 weeks at the screening visit.
3. Foot ulcer size is between 1 cm2 and 15 cm2
4. Ulcer graded I or II by Wagner grade, and extended to skin, tendon, and subcutaneous tissue.
5. Free of necrotic debris at target ulcer
6. Around ulcer area blood circulation should be secured to meet one of below criteria;

   * Blood vessels around the ulcer detected by Doppler Test
   * 0.7 < Ankle Brachial Index(ABI) < 1.3
   * Transcutaneous Oxygen Pressure, TcPO2 higher than 30 mmHg
7. Subject is able to give written informed consent prior to study start and to comply with the study requirements during study.

Exclusion Criteria:

1. Non-diabetic pathophysiologic ulcer.
2. The ulcer has increased or decreased in size by 30% or more during one week after the screening visit.
3. Subjects requiring intravenous (IV) antibiotics to treat infection.
4. Current evidence of infection including pus drainage from the wound site.
5. Subject has a glycated hemoglobin A1c (HbA1c) level of > 15%
6. Subject's blood sugar is > 450 mg/dl at postprandial.
7. Subjects with severe renal failure that cannot be managed by renal dialysis.
8. Subjects with severe hepatic deficiencies.
9. Subject is Human Immunodeficiency Virus (HIV) positive.
10. Subject who has allergic or hypersensitive reaction to bovine-derived proteins or fibrin glue.
11. Subject who is pregnant or breast-feeding.
12. Subjects who are unwilling to use an "effective" method of contraception during the study.
13. Subjects who have a clinically relevant history of alcohol or drugs abuse.
14. Subjects who are not able to understand the objective of this study or to comply with the study requirements.
15. Subjects who are considered to have a significant disease which can impact the study by investigator.
16. Subjects who are considered not suitable for the study by investigator.
17. Subjects who had had a history of surgery for malignant tumor within the last five years (except carcinoma in situ).
18. Subjects who are currently or are enrolled in another clinical study within 60 days of screening.
19. Subjects who have undergone wound treatments with growth factors, dermal substitutes, or other biological therapies within the last 30 days.
20. Subjects who are receiving oral or parenteral corticosteroids, immunosuppressive, or cytotoxic agents with unstable dose prior to 4 weeks from screening.
21. Subjects not comply with off-loading procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Proportions of subjects who achieved complete wound closure | During 12 weeks

SECONDARY OUTCOMES:
Time taken to complete wound closure between the two groups | During 12 weeks
Proportions of subjects who achieved complete wound closure | Follow up to 12 weeks
Proportions of subjects who achieved complete wound closure by the classification of Wagner Grade between the two groups | Follow up to 12 weeks
Change rates in wound size and depth compared to baseline between the two groups | During 12 weeks
  cm^2
Proportions of subjects who achieved complete wound closure at every visit by the classification of ulcer locations | Follow up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Kyu Han, MD. Ph D., Principal Investigator — Korea University Guro Hospital; Ki-Won Young, MD. Ph D., Principal Investigator — Eulji General Hospital; Junpyo Hong, MD. Ph D., Principal Investigator — Asan Medical Center; Donghyeok Shin, MD. Ph D., Principal Investigator — Konkuk University Medical Center; Junhyeong Kim, MD. Ph D., Principal Investigator — Keimyung University Dongsan Medical Center; Kang Chan, MD. Ph D., Principal Investigator — Chungnam National University Hospital; Hyungmin Hahn, MD. Ph D., Principal Investigator — Ajou University Medical Center; Changsik Park, MD. Ph D., Principal Investigator — Seoul National University Bundang Hospital; Youngkoo Lee, MD. Ph D., Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Korea University Kuro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided